CLINICAL TRIAL: NCT06372327
Title: Move Often eVery Day 2.0
Acronym: MOVD
Status: Enrolling by invitation | Phase: Not Applicable | Type: Interventional
Sponsor: Stanford University (Other)
Responsible Party: Principal Investigator, Marily Ann Oppezzo, Instructor of Medicine, Stanford Prevention Research Center, Stanford University
Allocation: Randomized | Model: Factorial | Masking: None | Purpose: Prevention
Other Study IDs: 73468
Record Dates: First submitted 2024-04-13; First posted 2024-04-18 (Actual); Last update posted 2025-08-03 (Actual); Status verified 2024-10

CONDITIONS: Exercise
Keywords: Sedentary Behavior
MeSH Terms: conditions — Motor Activity; Sedentary Behavior

STUDY DESIGN:
Intervention Model Description: This will be a 2 (Exercise snack number) x 2 (Exercise snack length) factorial design.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (4):
- 1 x 1 minute Exercise Snack / Day (Experimental): Participants will be assigned a daily goal of 1, 1-minute exercise snack to break up prolonged sitting.
  Interventions: Behavioral: Daily Exercise Snacks
- 1 x 4 Exercise Snack / Day (Experimental): Participants will be assigned a daily goal of 1, 4-minute exercise snack to break up prolonged sitting.
  Interventions: Behavioral: Daily Exercise Snacks
- 4x1 Exercise Snacks / Day (Experimental): Participants will be assigned a daily goal of 4, 1-minute exercise snack to break up prolonged sitting.
  Interventions: Behavioral: Daily Exercise Snacks
- 4x4 Exercise Snacks/Day (Experimental): Participants will be assigned a daily goal of 4, 4-minute exercise snack to break up prolonged sitting.
  Interventions: Behavioral: Daily Exercise Snacks

INTERVENTIONS:
Behavioral: Daily Exercise Snacks — Participants will be encouraged to break up prolonged sitting at work with brief, high-intensity exercise snacks of varying length / total number depending on condition assignment.

SUMMARY:
The purpose of this study is to assess a novel, widely-accessible intervention to both promote active breaks from work and improve cognitive and psychological performances at work in motivationally-accessible bouts. This will be done by interrupting prolonged sitting with 1-4 short (1-4 minutes), moderate-to-vigorous physical activity (MVPA) bouts with no equipment, and simple video-based instructions. The short bouts will be referred to as "exercise snacks." In this proposed exercise snacks intervention, investigators explicitly target a population with sedentary jobs due to the generalizability.

DETAILED DESCRIPTION:
Participants will answer a short 5-10-minute survey to determine eligibility. Eligible candidates will be invited to attend a 30-minute self-directed orientation session to provide a description of the consent form, study objectives and time commitments, the purpose of randomization, and the importance of completing follow-up assessments regardless of outcome. After the orientation sessions, interested and eligible individuals will be sent the e-consent form.

After participants consent to the study, they will be invited to take the baseline survey, and get assistance with study account set-ups (Garmin, GroupMe). Researchers will handle account set ups. Participants will be asked to download both apps and sign into the apps with the study provided accounts. Many individuals may have GroupMe accounts and will be asked to make a profile for their buddy chat with whatever name they prefer (able to hide their real name if preferred). Baseline measures will last for 2 weeks. And then the 6-week intervention will begin.

All consented participants will receive a 6-week intervention. The study is a 2x2 factorial design with 4 different group. We will be assessing the length of snacktivities (1 minute versus 4 minutes) as well as frequency of snacktivities through the day (1 per day versus 4 per day). Therefore, participants will be randomized into 4 groups: One 1-minute snacktivity per day, four 1-minute snacktivities per day, one 4-minute snacktivity per day, or four 4-minute snacktivities per day.

The intervention will consist of the following empirically supported components shown to promote engagement, adherence, and behavior change:

1. Self-monitoring of activity: Participants will be instructed to timestamp and track their snacktivities each day using their phone. Each participant will receive bracelets (1 or 4) that can used to track progress. For example, participants will be taught how they can move the bracelets from one arm to the other to act as a visual aid of how many snacktivities they have done each day.
2. Nightly reporting: Participants will be sent nightly texts to track progress on snacktivities as well as productivity, alertness, and physical energy.
3. Weekly progress reports and tailored feedback: Each week of completion the participant will get a report of their adherence to the protocol for that week and their goals for next week. Embedded in the progress report will be a link for an interactive action plan survey to plan next week's exercises; the action plan is personalized, and incorporates motivational interviewing and problem-solving strategies. Action planning has high acceptability and is identified as an effective behavioral technique that enhances self-monitoring.
4. Relatable modeling: Social modeling theory supports the use of relatable models representing the learner in behavior change and motivation. Dr. Oppezzo's previous work showed high acceptability when the exercise video models were representative of a diverse -body, -ethnicity, and -aged population. Each snacktivity instructional video will feature diverse models performing the moves in work clothes.
5. Barrier problem solving: At baseline, study team members will work with participants to identify a feasible, safe, and comfortably private workday location for performing the activity breaks.
6. Peer support: participants will be assigned a peer buddy who will act as a health-buddy motivational coach. This person will be in a private group-chat with their designated buddy (another participant) and our study account. The study account will monitor conversation and give motivational prompts, when needed, to boost conversation amongst the 2 buddies.

During the maintenance phase (after the intervention phase and lasting 6 months), participants will take part in booster sessions. The first 2 booster sessions will be completed every month, and the following 2 booster sessions will be completed every 6 weeks, following a scaffolded design to ease participants off of the program.

During the follow-up, investigators will collect behavioral data only via zoom. At the end of the study, we will conduct semi-structured interviews on study experience.

ELIGIBILITY:
Inclusion Criteria:

* Participants must be 30 years of age or older.
* English speaking
* Sedentary job with 90% of the work day sitting
* Not currently taking regular activity breaks at work

Exclusion Criteria:

* Yes to any Physical Activity Readiness Questionnaire questions or any condition where increased activity is contraindicated
* Currently doing another worksite physical activity intervention

Min Age: 30 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 40 (Estimated)
Dates: Start 2024-07-31 (Actual); Primary Completion 2026-07-01 (Estimated); Study Completion 2026-07-01 (Estimated)

PRIMARY OUTCOMES:
Number of self-reported exercise snack breaks at work at week 7 | Collected 1 work week at week 7 (the week after the 6 week intervention)
  For the post-test week after the 6 week intervention, participants will self-report the number of exercise snacks they do each day.
Number of self-reported exercise snack breaks at work at week 18 | collected 1 work week at week 18 (3 months after the intervention)
  For one week (at week 18) participants will self-report the number of exercise snacks they do each day.
Number of self-reported exercise snack breaks at work at week 30 during follow-up | collected 1 work week at week 30 (6 months after the intervention)
  For one week (at week 30) participants will self-report the number of exercise snacks they do each day.

SECONDARY OUTCOMES:
Liking of exercise snacks | at week 7, post test, immediately after 6 weeks of treatment
  5-point likert scale From not at all to extremely of how much did you like doing exercise snacks

CONTACTS AND LOCATIONS:
Overall Officials: Marily Oppezzo, PhD, Principal Investigator — Stanford University
Locations (1):
- Stanford University School of Medicine, Stanford, California, United States